CLINICAL TRIAL: NCT03475576
Title: Together in Line, the Power of Informal Care in Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Birgitte Schoenmakers, Professor Dr., KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Together in line - Cera
Record Dates: First submitted 2018-03-09; First posted 2018-03-23 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Quality of Life
Keywords: elderly; caregiving; needs; support

STUDY DESIGN:
Intervention Model Description: before and after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all participants (Other): The intervention, offered to the older civilians and their informal care groups will consist of a updated version of the 'Keuzewijzer'. This is a self-management tool which stimulates the communication within the informal care groups to make behaved choices concerning the care for the older civilian, taking into account the standards, values, concerns and needs of every informal caregiver and older civilian.
  Interventions: Other: Keuzewijzer

INTERVENTIONS:
Other: Keuzewijzer — The intervention, offered to the older civilians and their informal care groups will consist of a updated version of the 'Keuzewijzer'. This is a self-management tool which stimulates the communication within the informal care groups to make behaved choices concerning the care for the older civilian, taking into account the standards, values, concerns and needs of every informal caregiver and older civilian. The most important value of this intervention is the approachability and the structured, but adjusted manner of support, focused on the individual context of care with their specific needs.
  The 'Keuzewijzer' is an online tool whereby, in conversation with the informal care group and older civilian, the following aspects will be discussed in the context of the care for the older civilian: 1) analyzing the problem, 2) detection of possibilities or alternatives, 3) clarifying of motives and feelings and 4) weighting between values.

SUMMARY:
An aging population means an increase of the oldest part of the population, resulting from a change in demographic behavior and an increasing lifespan. The social networks are changing and the health care costs are rising. We know informal care of older civilians becomes more and more complex. A formal framework with a good communication to support informal caregivers is therefore essential in order to provide good care for a dependent older civilian.

Informal care is the support and assistance of a dependent person, outside the context of professional care or organized volunteering, but by one or more members from the immediate vicinity of the dependent1. The 'informal care group' is defined as follows: 'a group of two or more persons who together provide informal care to a dependent person, beyond the scope of professional care or organized volunteering, but as members of the immediate vicinity of the dependent'.

In this group, the different members contribute to the care process in an equitable but non-proportional manner. The dynamics in an informal care group are obviously different from those in a family where one central informal caregiver is responsible for the care of the ill relative: behind each individual of the informal care group, there is also a partner and/or children who influence the care motivations and accountability.

Sharing informal caregiving has important advantages. Firstly, individuals of the informal care group needs less time to fulfill specific caregiver tasks and have more time to cope with external stressors. Secondly, caregivers in group receive support from each other, which strengthens their self-efficacy. However, the involvement of more caregivers may also be a source of conflict.

This project aims to meet the needs of informal care groups of older civilians. An adjusted support for older civilians (≥70 years) and their informal care group will be achieved. We will focus on their needs, aimed to decrease the caregiver burden and increase the well-being of both older civilian and caregivers. This goal will be achieved by a better care planning and attempts to improve communication between older civilian, informal and professional caregivers, which we found in previous research as difficult and an important obstacle in concretize individual tailored support of the older civilian and caregivers.

DETAILED DESCRIPTION:
1. Study design The study has a before-and-after study design, the tailored support will be available for every informal care group and no older civilian will be excluded from an optimal care context, which is required by the social framework of this project. Therefore, no control group will be included in this study. The intervention consists of already existing support, although it is strengthened by means of a self-management tool, the 'Keuzewijzer', which helps the informal care group making specific choices with regard to tailored support, adjusted to their needs, norms and values. By a pre- and post-test, the effect of the intervention on the psychosocial well-being of the informal caregivers can be mapped out.
2. Study population 2.1. Study population definition In this study, informal care groups of older civilians will be included. These civilians will be 70 years or older and have to live independently at home in the Leuven region. The informal care groups consist of two or more relatives, friends or neighbors caring for the older civilian (≥70 years), beyond the scope of professional care or organized volunteering. There are no age restriction for the informal caregivers.

   2.2. Inclusion and exclusion criteria Both the older civilians and the informal caregiver give their written consent after being informed. Only civilians aged 70 years or older and their informal caregivers who have a thorough command of Dutch will be included. Older civilians with a formal diagnosis of dementia, too ill to participate or in a palliative phase be excluded.
3. Intervention The intervention, offered to the older civilians and their informal care groups will consist of an updated version of the 'Keuzewijzer', which has been developed in an earlier phase of the research project. This is a self-management tool which stimulates the communication within the informal care groups to make behaved choices concerning the care for the older civilian, taking into account the standards, values, concerns and needs of every informal caregiver and older civilian.

   The following aspects will be discussed in the context of the care for the older civilian: 1) analyzing the problem, 2) detection of possibilities or alternatives, 3) clarifying of motives and feelings and 4) weighting between values. The first purpose of this intervention is to develop a care planning focused on the older civilians with a clear distribution of tasks. The second purpose is to stimulate the communication between the informal caregivers and the older civilian, allowing timely adjustments in the care planning and preventing for caregiver burden.

   The intervention consist of the following parts: 1) introduction conversation, 2) Keuzewijzer and 3) follow-up conversation. In addition, an evaluation of the intervention takes place at the end of the intervention study (6 months).

   3.1. Introduction conversation During this conversation, a researcher will explain the dual purpose of the study, in which on the one hand the psychosocial well-being of the informal caregivers and the older civilian is mapped by means of the personal interviews and on the other hand, tailored support is offered through the intervention.

   The aim of this conversation consists of two aspects: 1.) providing information about the study and the informed consent and 2.) making the informal care group sensitive to its own care context and the concerns and needs that exist.

   3.2. Intervention The intervention consists, as explained earlier, of a self-management tool based on the 'Keuzewijzer'. Both the individual members of the informal care group and the older civilian must complete this online tool individually, preferably shortly after the introduction conversation. After completing the 'Keuzewijzer, the participants gets an overview of advice and referrals. Hereby, the informal care group gains insight into which existing support is available in response to their needs, concerns, values and standards. Direct contact can be made with the organizations involved and the tailored support can be started.

   The aim of the intervention is to strengthen existing support for informal caregivers and to tailor this support on the needs and concerns of the informal care groups.

   3.3. Finishing conversation and evaluation of the intervention After the intervention, the informal care group is offered a final conversation (6 months), in which the effect of the intervention will be discussed and the intervention itself will be evaluated. In addition, this conversation offers the opportunity to discuss and refer to any outstanding needs and concerns. A project employee will also guide this conversation.

   Together with the finishing conversation, the informal caregivers and the older civilian are given the opportunity to evaluate the intervention by means of a focus group.

   The aim of this conversation is to consider together with the informal care group 1) the effect of the intervention, 2) the possible concerns and needs to refer if necessary and 3) the intervention itself.
4. Data collection The study will take place over the period of 6 months with two measurement moments: within one month after including (baseline) and 6 months after inclusion. The informal care groups and the older civilians will be questioned individually through a web survey about their general everyday functioning and physical and psychosocial well-being. In addition, current support (apart from the study related support) focused on the older civilian or caregiver needs will be accurately recorded. This will allow to evaluate whether this contaminates the effect of the study intervention. When a caregiver or older civilian is unable to complete the questionnaire online, a paper version will be offered.

   4.1. Baseline data collection

   At the first measurement moment (baseline), data will be collected through online questionnaires. The questionnaires of both older civilian and caregiver will consist of the following parts:

   4.1.1. Informal caregiver
   * Background, functional status and caregiving The information about the background and functional status of the informal caregiver will comprise 1) socio-demographic information, e.g. age, living conditions, education and ethnicity and 2) physical well-being, like subjective health evaluation, visits to the GP and use of (prescribed and OTC) medication. The information about caregiving will comprise 1) type of caregiving tasks, 2) time investment 3) social and financial consequences of caregiving and 4) caregiving in group, e.g. division of tasks, communication, group cohesion and dynamics.
   * Psychosocial well-being

   Regarding the psychosocial well-being of the caregivers of the informal care group, the structured interviews will consist of the following questionnaires:
   * Zarit Burden Inventory The Zarit burden interview (ZBI), a self-report scale, is believed to be the most commonly used measure of caregiver burden. Bachner et al. showed that the ZBI was reliable across populations of caregivers and patients.
   * Geriatric Depression Scale The most commonly used scale for late-life depression is the geriatric depression scale (GDS). The 15-item GDS has been shown to have adequate sensitivity and specificity and to be significantly more accurate than the 30-item GDS.
   * State Trait Anxiety Inventory This subscale evaluates relatively stable aspects of anxiety, including general states of calmness, confidence and security. In this study, the Dutch version of the STAI will be used: The 'Zelf-Beoordelings Vragenlijst' (STAI-DY).
   * Spiritual resources & needs The spiritual resources and needs of the individuals of the informal care group and the older civilian will be questioned through open questions.

     * Support In this part of the structured interview, informal caregiver will be asked about the current formal and informal support and their knowledge about available support and information channels. The informal caregiver will also be asked about their role and experiences in the informal care group.

   4.1.2. Older civilians
   * Functioning The information about the functioning of the older civilians will comprise 1.) socio-demographic information, like age, living conditions, education and ethnicity, 2.) disease and treatment characteristics, 3.) activities of daily living (ADL, Barthel index) and 4.) instrumental activities of daily living (IADL, Lawton scale).
   * Psychosocial well-being Regarding the psychosocial well-being of the older civilians, the structured interviews will consist of the same questionnaires as for the informal caregivers, except the Zarit Burden Inventory. Besides, the loneliness of the older civilian will be measured. Loneliness is the subjective experience of social isolation and is associated with the well-being of community-dwelling older persons. Loneliness has been less well studied and may be less definable than depression or social support. But loneliness should certainly not be neglected as it has been shown that it is associated with adverse health consequences of older civilians. In the Netherlands, the loneliness scale of De Jong Gierveld and Kamphuis is generally used. As this scale has been developed in Dutch, has been used among older persons and has been proven to be a reliable and valid instrument that is robust to different data collecting modalities, this scale will be used.
   * Support In this part of the structured interview, the older civilian will be asked, like the informal caregiver, about the current (in)formal support and their knowledge about available support and information.

   4.2. Data collection during follow-up The data collection during follow-up will also take place online through a web survey. The Zarit Burden Inventory (ZBI-12 items) and the Geriatric Depression Scale (GDS-15 items) will be included in the follow-up interview of the informal caregiver, examine changes in their psychosocial well-being over time. Besides, the follow-up interviews also include questions about their physical well-being, support, functioning of the informal care group and socio-demographics. The spiritual well-being, coping and state anxiety of the informal caregiver are considered to remain stable over 6 months, so these items will not be questioned again. The follow-up interview of the older civilian will include the Geriatric Depression Scale (GDS-15 items), Activities of Daily Living (ADL, Barthel index) and the Instrumental Activities of Daily Living (IADL, Lawton IADL scale), besides socio-demographic questions.
5. Statistical analysis Standard statistical analyses will be used for describing the characteristics of the older civilian and informal care group at baseline and during follow-up.

When applicable more complex statistical methods will be used. For example, odds ratios and 95% confidence intervals for the different outcome parameters (e.g. functional status, physical and psycho-social well-being) will be estimated using multivariable logistic regression models.

ELIGIBILITY:
Inclusion Criteria:

* Both the older civilians and the informal caregiver give their written consent after being informed.
* Only civilians aged 70 years or older and their informal caregivers will be included.
* Only civilians and their informal caregivers who have a thorough command of Dutch will be included.

Exclusion Criteria:

* Older civilians with a formal diagnosis of dementia
* too ill to participate
* in a palliative phase

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
caregiver burden | 6 months
  The Zarit burden interview (ZBI), a self-report scale, is believed to be the most commonly used measure of caregiver burden. Initially the ZBI was developed to measure strain associated with the care of community-dwelling persons with Alzheimer disease, but Bachner et al. showed that the ZBI was reliable across populations of caregivers and patients.
  The ZBI was used to assess the subjective burden experienced by an informal caregiver. For this study an adjusted 12 item ZBI, derived from the QUALIDEM Project, was chosen. The answers are never, rarely, sometimes, quite frequently and nearly always (scored from 0 to 4). The sum was taken over all the questions (range 0-48) and the caregiver was assigned to a category of severe or high burden if the score was 17 or higher. The standard ZBI-12 of Bedard et al. has shown a high correlation with the full ZBI ranging from 0.92 to 0.97 (p=0.001).
depressive complaints | 6 months
  Geriatric Depression Scale: The most commonly used scale for late-life depression is the geriatric depression scale (GDS).
  The GDS is an instrument to measure depressive complaints specifically in an older population. However, Covinsky et al. has also used it to screen for caregiver depression. The short version will be used, which consists of 15 yes or no questions. The scores are summed range 0-15 and the participant is categorised as having depressive complaints when he or she scores five or higher. The 15-item GDS has been shown to have adequate sensitivity and specificity and to be significantly more accurate than the 30-item GDS.

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Schoenmakers, PhD, Principal Investigator — ACHG
Locations (1):
- ACHG, Leuven, Belgium